CLINICAL TRIAL: NCT00454610
Title: Family Lifestyle Overweight Prevention Program: Evaluation of a Weight Management Program for Mexican American Youth
Brief Title: Family Lifestyle Overweight Prevention Program
Acronym: FLOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, John P. Foreyt, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H15671
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Overweight; Obesity
Keywords: Pediatric; Overweight; Obesity; Intervention; Prevention; Mexican American
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: FLOW
Behavioral: SelfHelp

SUMMARY:
The purpose of the study was to design a weight management program for Mexican American youth and to determine the effectiveness of the program for weight management compared to a self help program.

1. At the end of 6 months, individuals randomly assigned to Intensive Intervention (II) (instructor/trainer led intervention) will lose more weight than individuals assigned to Self Help (SH) only.
2. At the end of 1 year, individuals randomly assigned to II will maintain their weight losses better than individuals assigned to SH.

Secondary hypotheses will include examination of main effects and interactions at the end of 6 months with the following secondary dependent measures: treatment adherence (e.g., attendance, food diaries, exercise diaries), blood levels, changes in percent body fat, overall psychological functioning (PEDS-QL 4.0), and eating behaviors as assessed by food frequency checklists.

DETAILED DESCRIPTION:
The overall objective of this study is to compare the effectiveness of a behavioral, family-based weight management program and a self-help only group for the prevention of obesity in adolescents. The treatments are; Self Help(SH) Instructions to follow a 12-week self help manual for healthy eating and increased physical activity; Intensive Intervention (II) 12 Weeks of daily and 7 Monthly sessions consisting of nutrition instruction, physical activity training, and behavior modification instruction. One hundred (BMI-for-age = 85th - 97.5th % or parent BMI > 25) adolescent males and females will be recruited into the study and randomly assigned to SH) Instructions to follow the self help manual for healthy eating and increased physical activity; II) 12 Weeks daily and 7 Monthly sessions consisting of nutrition instruction, physical activity training, and behavior modification instruction for one year. Participants will receive final measurements at the end of year 1 and intermediate evaluations at month 6. Given that the interventions decline in intensity and frequency after 3 months, the 1 year assessments will help evaluate which treatment was most effective in maintaining weight losses with minimal contact.

SH will consist of participants being instructed to follow a 12-week parent/child based self help book for weight loss, but they will not receive any active intervention. The manual (TRIM Kids, Sothern, von Almen, & Schumacher, 2001) that the families will follow is a treatment program which uses a family-based, behavioral intervention that focuses on diet and exercise with instructions and guidelines designed to assist the family in maintaining weight losses. II will consist of 12 Weeks of daily and 7 Monthly sessions consisting of nutrition instruction, physical activity training, and behavior modification instruction over the 1-year period. Body mass index (BMI), blood analyses (i.e. cholesterol, triglycerides, insulin, glucose, C-reactive protein, mono-unsaturated fatty acids, and inflammatory cytokines), analysis of eating and exercise behavior, and eating and exercise self-efficacy measures will be taken throughout the study. The focus of this study is to evaluate the effectiveness of an active, behaviorally designed intervention for the prevention of adult obesity.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the 6th or 7th grade at the target school.
* Parent consent and child assent to participate.

Exclusion Criteria:

* Taking medications for weight control.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2005-01; Study Completion 2007-03

PRIMARY OUTCOMES:
standardized body mass index (zbmi)

SECONDARY OUTCOMES:
blood levels,
changes in percent body fat,
overall psychological functioning
eating behaviors

CONTACTS AND LOCATIONS:
Overall Officials: John P Foreyt, Ph.D., Principal Investigator — Baylor College of Medicine

REFERENCES:
- [Background] Tyler C, Johnston CA, Fullerton G, Foreyt JP. Reduced quality of life in very overweight Mexican American adolescents. J Adolesc Health. 2007 Apr;40(4):366-8. doi: 10.1016/j.jadohealth.2006.10.015. Epub 2007 Feb 5. PMID 17367735
- [Result] Johnston CA, Tyler C, Fullerton G, Poston WS, Haddock CK, McFarlin B, Reeves RS, Foreyt JP. Results of an intensive school-based weight loss program with overweight Mexican American children. Int J Pediatr Obes. 2007;2(3):144-52. doi: 10.1080/17477160701305864. PMID 17999280
- [Result] Fullerton G, Tyler C, Johnston CA, Vincent JP, Harris GE, Foreyt JP. Quality of life in Mexican-American children following a weight management program. Obesity (Silver Spring). 2007 Nov;15(11):2553-6. doi: 10.1038/oby.2007.306. PMID 18070745
- [Derived] Johnston CA, Palcic JL, Tyler C, Stansberry S, Reeves RS, Foreyt JP. Increasing vegetable intake in Mexican-American youth: a randomized controlled trial. J Am Diet Assoc. 2011 May;111(5):716-20. doi: 10.1016/j.jada.2011.02.006. PMID 21515118
- [Derived] Johnston CA, Tyler C, Fullerton G, McFarlin BK, Poston WS, Haddock CK, Reeves RS, Foreyt JP. Effects of a school-based weight maintenance program for Mexican-American children: results at 2 years. Obesity (Silver Spring). 2010 Mar;18(3):542-7. doi: 10.1038/oby.2009.241. Epub 2009 Aug 6. PMID 19661957
- [Derived] Johnston CA, Tyler C, McFarlin BK, Poston WS, Haddock CK, Reeves R, Foreyt JP. Weight loss in overweight Mexican American children: a randomized, controlled trial. Pediatrics. 2007 Dec;120(6):e1450-7. doi: 10.1542/peds.2006-3321. PMID 18055663